CLINICAL TRIAL: NCT03164278
Title: Studying the Effectiveness of Remote Training
Brief Title: Effectiveness of Web-Based Training (SERT)
Acronym: SERT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Boninger, Professor and UPMC Endowed Vice Chair for Research, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY19020341; 90SI5014-01-00 (Other Grant/Funding Number: U.S. Department of Health and Human Services)
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Remote Transfer Training Program
Keywords: Wheelchair; Biomechanics; Transfer; Participation; Training

STUDY DESIGN:
Intervention Model Description: This is a randomized single blind study.
Masking Description: Subjects will be choose to be in one of three groups: one group will receive transfer training immediately with no follow up, one group will receive the transfer training immediate with a 1 month & 6 month follow up, and one group that will be randomized to either receive the transfer training immediately or to receive the transfer training after a 6 month wait (with follow ups).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate Training (no follow up) (Experimental): Individuals may decide to participate in the research study training program, but not in any follow up questionnaires. This group will have immediate access to the independent transfer training materials. They will complete data collection measures embedded in the transfer training program, including demographics, Online Learning Readiness Scale (OLRS), Moorong Self Efficacy Scale (MSES), Patient Reported Outcome Measurement Information System (PROMIS), Transfer Assessment Instrument Questionnaire (TAI-Q), and the Wheelchair User Shoulder Pain Index (WUSPI).
  Interventions: Behavioral: Independent Transfer Training
- Immediate Training (with follow up) (Experimental): Individuals may decide to participate in the research study, but do not want to be randomized. After consent is obtained, these individuals will be directed immediately to the baseline questionnaires (see above) before and after the independent transfer training. Participants may also be asked to complete a user satisfaction survey.
  Interventions: Behavioral: Independent Transfer Training
- Randomized Training (Experimental): Individuals may decide to participate in the research study and agree to be randomized. These individuals will be immediately randomized into an immediate or a wait list control group. The immediate will receive the independent transfer training program after completing the baseline questionnaires. The wait list control group will wait approximately 6 months before receiving the independent transfer training program.
  Interventions: Behavioral: Independent Transfer Training

INTERVENTIONS:
Behavioral: Independent Transfer Training — Independent Transfer Training Program: ITTP training starts with an overview and self-evaluation using the transfer assessment instrument questionnaire (TAI-Q) followed by three core modules: wheelchair setup, body setup, and flight/landing. Wheelchair setup includes factors such as the angle and distance of the wheelchair to the transfer surface, removing barriers, applying the brakes, and height of the transfer. Body setup involves positioning one's body for an optimal transfer and covers foot, hip, arm and hand positions. Flight/landing discusses how to achieve a smooth and controlled transfer, the head-hips relationship, use of transfer device, and safe landing.

SUMMARY:
The objective of this research study is to assess the effectiveness of an independent transfer training program (ITTP), and to determine methods which may increase overall success of an online training program.

DETAILED DESCRIPTION:
Up to 200 individuals will be recruited for this research study. Investigators will recruit individuals who use a wheelchair for the majority of their mobility (over 40 hours per week), have the ability to transfer independently (may use equipment like sliding boards), use a seated pivot to transfer, and speak English as a primary a language. This study will be accessed entirely online and participation is expected to last approximately one year. Subjects will be randomized into three groups; one group that will receive transfer training immediately with no follow up, one group that will receive the transfer training immediately with 1 month and 6 month follow up, and one group that will receive the transfer training after 6 months. The transfer training program itself will take approximately 1 hour to complete.

After obtaining informed consent, participants in the first two groups will complete baseline questionnaires. They will then receive the transfer training program.

Participants in the third group (a wait-list control group) will complete the baseline questionnaires and be contacted one month later to complete a transfer assessment instrument questionnaire. They will then wait 5 months. After this period, participants will complete the baseline questionnaires a second time, and then receive the transfer training.

After completing the transfer training, all groups will be contacted immediately post training to complete additional questionnaires to assess the effectiveness of the remote transfer training program. Participants in the 2nd and 3rd group will be contacted 1 month and 6 months post-training to complete additional questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Utilize a wheelchair for the majority of mobility (over 40 hours per week).
2. Ability to transfer independently (may use equipment like sliding boards).
3. Use of seated pivot transfer
4. Speak English as a primary a language

Exclusion Criteria:

1. Pain prohibiting transfers
2. Active use of the lower limb muscles during transfers
3. Current or recent history (last 3 months) of pressure sores

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-12-04 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Transfer Assessment Instrument Questionnaires (TAI-Q) | This measure is collected at baseline, pre- training, during the training, as well as at the 1 month and 6 month follow ups.
  We will assess the mathematical difference in assessments from baseline to follow-up.

SECONDARY OUTCOMES:
Change in Wheelchair Users Shoulder Pain Index (WUSPI) | This measure is collected pre- training, as well as at 6 month follow up.
  We will assess the mathematical difference in assessments from baseline to follow-up.
Change in Patient Reported Outcomes Measurement Information System: Physical Function with Mobility Aid | This measure is collected pre-training and at the 6 month follow up.
  We will assess the mathematical difference in assessments from baseline to follow-up.
Change in Patient Reported Outcomes Measurement Information System: Satisfaction with Social Roles & Activities | This measure is collected pre-training and at the 6 month follow up.
  We will assess the mathematical difference in assessments from baseline to follow-up.
Change in Patient Reported Outcomes Measurement Information System: Ability to Participate in Social Roles and Activities | This measure is collected pre-training and at the 6 month follow up.
  We will assess the mathematical difference in assessments from baseline to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Boninger, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The American Institutes for Research (AIR) will have access to the de-identified questionnaire data and will participate in the private Facebook forum. Requests from AIR to access the data will be made to the Principal Investigator.
Time Frame: Supporting information will be shared with collaborators per data sharing agreement guidelines.
Access Criteria: Contact a study team member for access criteria.

REFERENCES:
- [Derived] Rigot SK, DiGiovine KM, Boninger ML, Hibbs R, Smith I, Worobey LA. Effectiveness of a Web-Based Direct-to-User Transfer Training Program: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2022 Apr;103(4):807-815.e1. doi: 10.1016/j.apmr.2021.05.007. Epub 2021 Jun 4. PMID 34090854